CLINICAL TRIAL: NCT03572231
Title: A Prospective, Non-interventional, Registry Study of Patients Initiating Pharmacologic Therapy for Overactive Bladder in Taiwan, Korea and China
Brief Title: A Registry Study of Patients Initiating a Course of Drug Therapy for Overactive Bladder in Taiwan, Korea and China
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Singapore Pte. Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 178-MA-3146
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Overactive Bladder (OAB)
Keywords: Betmiga; OAB; YM178; Overactive Bladder; mirabegron
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — mirabegron; darifenacin; imidafenacin; Tolterodine Tartrate; oxybutynin; trospium chloride; fesoterodine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mirabegron: Participants will commence the OAB treatment with mirabegron that is prescribed by a physician in routine clinical practice.
  Interventions: Drug: mirabegron
- Antimuscarinics: Participants will commence the OAB treatment with one of the following antimuscarinics: solifenacin, darifenacin, imidafenacin, tolterodine, oxybutynin, trospium, fesoterodine or propiverine. The antimuscarinic is prescribed by a physician in routine clinical practice.
  Interventions: Device: solifenacin; Drug: darifenacin; Drug: imidafenacin; Drug: tolterodine; Drug: oxybutynin; Drug: trospium; Drug: fesoterodine; Device: propiverine

INTERVENTIONS:
Drug: mirabegron — oral
  Other Names: YM178; Betmiga
  Groups: mirabegron
Device: solifenacin — oral
  Other Names: YM905; Vesicare
  Groups: Antimuscarinics
Drug: darifenacin — oral
  Groups: Antimuscarinics
Drug: imidafenacin — oral
  Groups: Antimuscarinics
Drug: tolterodine — oral
  Groups: Antimuscarinics
Drug: oxybutynin — oral
  Groups: Antimuscarinics
Drug: trospium — oral
  Groups: Antimuscarinics
Drug: fesoterodine — oral
  Groups: Antimuscarinics
Device: propiverine — oral
  Groups: Antimuscarinics

SUMMARY:
The purpose of this study is to observe and describe treatment patterns, like Overactive Bladder (OAB) treatment discontinuation, switching to other therapies and persistence of OAB therapies in routine clinical practice.

This study will also evaluate effectiveness of OAB therapies in routine clinical practice; identify factors associated with effectiveness and persistence of pharmacologic therapies in OAB participants; evaluate the Quality of Life (QoL) and treatment satisfaction of OAB therapies; as well as evaluate health care resource utilization (HCRU) and understand adverse events (AEs), serious adverse events (SAEs) and adverse drug reactions (ADRs) associated with OAB therapies.

DETAILED DESCRIPTION:
This is an observational registry study and will not provide or recommend any treatment; all decisions regarding treatment are made at the sole discretion of the treating physician in accordance with the treating physician's usual practices and all eligible participants will be enrolled in a certain timeframe. OAB participants enrolled in the study will be categorized into one of two treatment groups, but the study does not plan to compare the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with OAB symptoms (with or without urgency incontinence) with symptoms for at least three months prior to study enrollment.
* About to initiate monotherapy of mirabegron or any antimuscarinics therapy for OAB symptoms, prescribed as part of routine clinical practice, which maybe the first course of any treatment for OAB, lapsed of treatment, or switching from one drug to another.

Exclusion Criteria:

* Currently receiving more than one medication (including Chinese herbal medicine) for OAB.
* Current participation in clinical trials of OAB.
* Have undergone surgery for OAB in the past.
* Mixed incontinence where stress incontinence is the predominant form.
* OAB has been treated with onabotulinum toxin A, sacral neuromodulation, percutaneous tibial nerve stimulation, external beam radiation (XRT), stents, surgery, or intermittent catheterization prior to or at time of enrollment.
* At risk of Acute Urinary Retention (AUR).
* Neurologic conditions associated with OAB symptoms.
* Hypersensitivity and contraindication(s) to mirabegron and antimuscarinics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and/or female adult OAB patients, whose physicians have decided to start OAB drug therapy in routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 805 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Time from treatment initiation to discontinuation of Overactive Bladder (OAB) therapy | Up to 26 weeks
  Discontinuation will include participants who discontinue mirabegron or antimuscarinics for more than 30 days (defined as the day after the last day of the prior supply to the next dispensing date).
Time from treatment initiation to switching to another OAB therapy or dose | Up to 26 weeks
  Switching will be defined as a subset of initial mirabegron or antimuscarinics discontinuers who initiated another/different therapy(ies) within the follow-up period or within 30 days of being prescribed the first treatment. Change of treatment to another formulation of the same drug type under the same dosage will not be considered as switching.
Proportion of participants who discontinue OAB treatment | Up to 26 weeks
  Discontinuation will include participants who discontinue mirabegron or antimuscarinics for more than 30 days (defined as the day after the last day of the prior supply to the next dispensing date).
Proportion of participants who switch to another treatment or dose | Up to 26 weeks
  Switching will be defined as a subset of initial mirabegron or antimuscarinics discontinuers who initiated another/different therapy(ies) within the follow-up period or within 30 days of being prescribed the first treatment. Change of treatment to another formulation of the same drug type under the same dosage will not be considered as switching.

SECONDARY OUTCOMES:
Change from baseline in Overactive Bladder Questionnaire-Short Form (OAB-Q-SF) score | Baseline, weeks 10-14 and weeks 22-26
  Overactive Bladder Questionnaire-Short Form (OAB-Q-SF) is a participant-reported instrument consisting of 19 items that assess the degree to which a participant is bothered by OAB symptoms, and the degree of impact of OAB symptoms on daily life. Participants rate each item using a 6-point Likert Scale ranging from "Not at all" to "A very great deal" for the symptom bother items and "none of the time" to "All of the time" for the Health Related Quality of Life (HRQL) items.
Change from baseline in Bladder Assessment Tool (BAT) score | Baseline, weeks 10-14 and weeks 22-26
  Bladder Assessment Tool (BAT) is a participant-reported instrument consisting of 17 questions regarding the symptoms, bothering, impacts and treatment satisfaction in the past 7 days. Scores range from 0 to 88, a reduction in BAT score indicates an improvement.
Change from baseline in Overactive Bladder Symptom Scores (OABSS) score | Baseline, weeks 10-14 and weeks 22-26
  Overactive Bladder Symptom Scores (OABSS) is a participant-reported instrument consisting of 4 questions regarding daytime frequency, nocturia, urgency, and urgency incontinence; evaluates relevant symptoms from the participant's viewpoint. Scores range from 0 to 15 with a lower score indicating a mild presentation of overactive bladder syndrome and a higher score indicating moderate to severe presentation of overactive bladder syndrome.
Change from baseline in Treatment Satisfaction-Visual Analog Scale (TS-VAS) score | Baseline, weeks 10-14 and weeks 22-26
  Treatment Satisfaction-Visual Analog Scale (TS-VAS) is a quantitative instrument assessing participant improvement in participants with OAB. A score of 10 on the TS-VAS indicates complete satisfaction, whereas a positive change from baseline indicates improvement.
Identify factors associated with the effectiveness and persistence of a pharmacologic therapy for an OAB participant: Demographic Information | Baseline (up to Day 0)
  Demographic information will be collected from participants for analysis.
Identify factors associated with the effectiveness and persistence of a pharmacologic therapy for an OAB participant: OAB Medical History | Baseline (up to Day 0)
  OAB medical history will be collected from participants for analysis.
Identify factors associated with the effectiveness and persistence of a pharmacologic therapy for an OAB participant: History of prior drug treatment for OAB | Baseline (up to Day 0)
  History of prior drug treatment for OAB will be collected from participants for analysis.
Identify factors associated with the effectiveness and persistence of a pharmacologic therapy for an OAB participant: Medical history | Baseline (up to Day 0)
  Medical history will be collected from participants for analysis.
Identify factors associated with the effectiveness and persistence of a pharmacologic therapy for an OAB participant: Concomitant medication information | Up to 26 weeks
  Concomitant medication will be collected from participants for analysis.
Identify factors associated with the effectiveness and persistence of a pharmacologic therapy for an OAB participant: Concomitant medical conditions | Up to 26 weeks
  Participants medical history will be collected from participants for analysis.
Health Care Resource Utilization (HCRU) related to the management of OAB | Up to 26 weeks
  Participant information will be collected by the investigator or designee via the Healthcare Resource Utilization (HCRU) Worksheet at each visit and the data will be retrieved electronically via the electronic case report form (eCRF). The HCRU worksheet consists of 7 questions related to the participants history and treatment of OAB.
Safety assessed by Adverse Events (AEs) | Up to 26 weeks
  An AE is any untoward medical occurrence in a patient or clinical study patient administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a product, whether or not considered related to the product. Pre-existing conditions that worsen during a study are to be reported as AEs.
Safety assessed by Serious Adverse Events (SAEs) | Up to 26 weeks
  Adverse event (AE) is considered "serious" if the investigator or sponsor view any of the following outcomes: Death, life-threatening, persistent or significant disability/incapacity, congenital anomaly or birth defect, hospitalization, or medically important event.
Safety assessed by Adverse Drug Reaction (ADR) | Up to 26 weeks
  An ADR is defined as any noxious and unintended response associated with the use of a drug in humans, at any dose, where a causal relationship (drug-event) is at least a reasonable possibility.

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Singapore Pte. Ltd.
Locations (15):
- South Korea (9):
  - Site KR410008, Daejeon
  - Site KR410009, Incheon
  - Site KR410005, Kangam
  - Site KR410001, Seoul
  - Site KR410002, Seoul
  - Site KR410003, Seoul
  - Site KR410006, Seoul
  - Site KR410007, Seoul
  - Site KR410004, Suwon
- Taiwan (6):
  - Site TW158001, Hualien City
  - Site TW158003, Kaohsiung City
  - Site TW158006, Kaohsiung City
  - Site TW158002, Taichung
  - Site TW158004, Taipei
  - Site TW158005, Taoyuan

REFERENCES:
- [Derived] Oh SJ, Cho ST, Kuo HC, Chou EC, Hsu YC, Lee KS, Hadi F, Song Y, Sumarsono B. Treatment Patterns with Mirabegron and Antimuscarinics for Overactive Bladder: A Prospective, Registry Study in Taiwan and South Korea (FAITH). Adv Ther. 2024 Apr;41(4):1652-1671. doi: 10.1007/s12325-024-02784-2. Epub 2024 Mar 2. PMID 38430402
- [Derived] Hadi F, Sumarsono B, Lee KS, Oh SJ, Cho ST, Hsu YC, Rasner P, Jenkins C, Fisher H. A treatment prediction strategy for overactive bladder using a machine learning algorithm that utilized data from the FAITH study. Neurourol Urodyn. 2023 Aug;42(6):1227-1237. doi: 10.1002/nau.25190. Epub 2023 May 6. PMID 37148497